CLINICAL TRIAL: NCT00471601
Title: Measuring Patient Expectations for Breast Reconstruction: Development and Validation of a Patient-Reported Outcomes Instrument
Brief Title: Development of a Questionnaire to Evaluate Patient Expectations for Breast Reconstruction in Women With Breast Cancer or Other Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); McMaster University (Other); University College, London (Other); The New School for Social Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-024; P30CA008748 (NIH); MSKCC-07024
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Psychiatric Rehabilitation

ARMS (1):
- Interviews/Questionnaires (Experimental): The primary intervention in part 1 includes the interview for item generation with 50 women and the pilot-testing with a separate group of n = 30 women. The primary intervention in part 2 and 3 is the administration of the questionnaire. In part 3, along with the questionnaire being developed, the Body Image Scale (BIS), the Life Orientation Test-Revised (LOT-R), and the upcoming MSKCC BREAST-Q will be given to determine convergent and discriminant construct validity. No other therapeutic or diagnostic agents will be administered.
  Interventions: Behavioral: counseling intervention; Behavioral: questionnaire administration; Behavioral: psychosocial assessment and care; Behavioral: quality-of-life assessment

INTERVENTIONS:
Behavioral: counseling intervention
Behavioral: questionnaire administration
Behavioral: psychosocial assessment and care
Behavioral: quality-of-life assessment

SUMMARY:
RATIONALE: A questionnaire that evaluates a patient's expectations about breast reconstruction surgery may help doctors improve patient education before surgery and increase patient satisfaction after surgery.

PURPOSE: This clinical trial is developing a questionnaire to evaluate patient expectations for breast reconstruction in women with breast cancer or other conditions.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and validate a questionnaire to evaluate preoperative expectations about breast reconstruction in women with breast cancer or other conditions.
* Determine variations in expectations related to patient characteristics.
* Develop educational modules to help patients understand realistic outcomes.
* Identify patient groups at risk for dissatisfaction.

OUTLINE: This is a 3-part study.

* Part 1 (first 80 patients): Both preoperative and postoperative patients (50 patients total) undergo an interview by a research study assistant about their expectations for breast reconstructive surgery. Some of these patients will also complete a pilot version of a questionnaire about their expectations for breast reconstructive surgery (30 patients total).
* Part 2 (next 200 patients): Preoperative patients complete questionnaires (the preliminary questionnaire developed after part 1 and the MSKCC BREAST-Q [Reconstruction Module]) about their expectations for breast reconstructive surgery after patient education about breast reconstructive surgery. Some of these patients (100 patients) also complete the Brief Cope addressing emotional expression and emotional processing styles of coping, Impact of Events Scale, and Life Orientation Test-Revised (LOT-R) questionnaires.
* Part 3 (final 200 patients): Preoperative patients complete a questionnaire (final questionnaire developed after part 2) about their expectations for breast reconstructive surgery after patient education about breast reconstruction and once after surgery. Patients also complete the Breast Reconstruction Outcomes Questionnaire (MSKCC BREAST-Q) once before surgery (after patient education) and once after surgery measuring patient satisfaction and quality of life. A small group of patients complete the Body Image Scale (BIS) and the LOT-R addressing body image, sexuality, personal well-being, and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age > or = to 18 to 75 years.
* Patients who are presenting for consultation about breast reconstruction

Exclusion Criteria:

* Inability to speak or understanding English
* Inability to provide meaningful informed consent due to physical, cognitive, or psychiatric disability.
* Prior breast reconstruction surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2007-03-13 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Item reduction | 2 years
Psychometric evaluation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McCarthy, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Peter G. Cordeiro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (2):
  - New School for Social Research, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario, Canada
- University College of London Hospitals, London, England, United Kingdom

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm